CLINICAL TRIAL: NCT02624518
Title: 68Ga-RM2 PET/MRI in the Evaluation of Patients With Biochemical Recurrence of Prostate Cancer and Non-contributory CT Scans
Brief Title: 68Ga-RM2 PET/MRI in Biochemically Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Principal Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-35155; NCI-2015-01993 (Other: NCI); PROS0074 (Other: Stanford Cancer Institute)
Record Dates: First submitted 2015-11-30; First posted 2015-12-08 (Estimated); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — BAY 86-7548; Gallium; Receptors, Bombesin; 68Ga-bombesin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (68Ga-RM2 PET/MRI) (Experimental): Patients receive 68Ga-RM2 IV and beginning 45 minutes later undergoing PET/MRI scan. The 68Ga-RM2 PET/MRI may be repeated at the completion of treatment to evaluate response to therapy, if requested by the treating physician. Imaging with PET/MRI is the intervention.
  Interventions: Drug: 68Ga-RM2; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: 68Ga-RM2 — Imaging with PET/MRI
  Other Names: Gallium (68Ga)-labeled gastrin-releasing peptide receptor (GRPr) antagonist; 68Ga-DOTA RM2; BAY 86-7548; 68Ga-Bombesin; DOT-bombesin
Procedure: Magnetic Resonance Imaging — Imaging with 68Ga-RM2 PET/MRI
  Other Names: Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI
Procedure: Positron Emission Tomography — Imaging with 68Ga-RM2 PET/MRI
  Other Names: PET

SUMMARY:
Prostate cancer (PC) remains the most-common non-cutaneous cancer diagnosed in American males, accounting for an estimated 174,560 estimated new cases and 31,620 estimated deaths in 2019. Up to 40% of the patients with prostate cancer develop biochemical recurrence within 10 years after initial treatment. Usually an increase of the prostate-specific antigen (PSA) llevel precedes a clinically detectable recurrence by months to years, and this is currently used as a screening test before and subsequent to treatment. However, disease advancement can be local, regional or systemic, and each has significantly different approaches to disease management. Unfortunately, PSA level does not differentiate between these disease stages.

This phase 2-3 study explores the utility of radiolabel 68Ga-RM2, a 68-gallium (68Ga)-labeled gastrin-releasing peptide receptor (GRPr) antagonist, for positron emission tomography (PET) / magnetic resonance imaging (MRI) (collectively, PET/MRI) as a potential tool to help discriminate between disease stages in participants after treatment with surgery or radiation, who present persistently elevated PSA levels (ie, may have prostate cancer), but were negative for cancer with a diagnostic regular medical care computed tomography (CT) scan

68Ga-RM2 (BAY86-7548) is also identified as a synthetic bombesin receptor antagonist. PET/MRI is the collective result of 2 scan processes (PET and MRI ) conducted during the same scan procedure (ie, a combined scan). After a regular medical care computed tomography (CT) scan, participants will be scanned with 68Ga-RM2 PET/MRI scan procedure. PET/MRI is used to assess the location, size, and metabolic activity of a suspected tumor.

The 68Ga-RM2 radiolabel consisted of a ligand (the synthetic bombesin receptor antagonist) and the radioisotope 68Ga. The RM2 ligand targets gastrin-releasing peptide receptors (GRPr), commonly expressed by prostate cancer cells, and the radioisotope distinguishes those cells from the background. The criteria for scan "positivity" will be, when compared to background level of the liver (control), the 68Ga signal is stronger (positive - malignant) or weaker (negative - benign).

This study will assess how well 68Ga-RM2 works in detecting prostate cancer in patients with

68Ga-RM2 PET/MRI may be able to see smaller tumors than the standard of care contrast-enhanced CT or MRI scan.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Evaluate 68Ga-RM2 as the radiolabel for PET/MRI scans used for detection of recurrent prostate cancer after initial therapy in patients with elevated prostate-specific antigen (PSA) and non-contributory computed tomography (CT).

OUTLINE:

Patients receive 68Ga-RM2 intravenously (IV) and beginning 45 minutes later undergoing PET/MRI scan. The 68Ga-RM2 PET/MRI may be repeated at the completion of treatment to evaluate response to therapy, if requested by the treating physician.

After completion of study, patients are followed up at 24 to 48 hours and then at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma
* Rising PSA after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy

  * Post radical prostatectomy (RP) - American Urological Association (AUA) recommendation

    * PSA greater than 0.2 ng/mL measured 6-13 weeks after RP
    * Confirmatory persistent PSA greater than 0.2 ng/mL
  * Post-radiation therapy - American Society for Therapeutic Radiology and Oncology (ASTRO)-Phoenix consensus definition

    * Nadir plus (+) greater than or equal to 2 ng/mL rise in PSA
* No evidence of metastatic disease on conventional imaging, including a negative bone scan for skeletal metastasis and negative contrast-enhanced CT
* Able to provide written consent
* Karnofsky performance status of >= 50 (or Eastern Cooperative Oncology Group [ECOG]/World Health Organization [WHO] equivalent)

Exclusion Criteria:

* Unable to provide informed consent
* Inability to lie still for the entire imaging time
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the investigator, may significantly interfere with study compliance
* Metallic implants

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2022-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baratto L, Song H, Duan H, Hatami N, Bagshaw HP, Buyyounouski M, Hancock S, Shah S, Srinivas S, Swift P, Moradi F, Davidzon G, Iagaru A. PSMA- and GRPR-Targeted PET: Results from 50 Patients with Biochemically Recurrent Prostate Cancer. J Nucl Med. 2021 Nov;62(11):1545-1549. doi: 10.2967/jnumed.120.259630. Epub 2021 Mar 5. PMID 33674398
- [Result] Baratto L, Duan H, Laudicella R, Toriihara A, Hatami N, Ferri V, Iagaru A. Physiological 68Ga-RM2 uptake in patients with biochemically recurrent prostate cancer: an atlas of semi-quantitative measurements. Eur J Nucl Med Mol Imaging. 2020 Jan;47(1):115-122. doi: 10.1007/s00259-019-04503-4. Epub 2019 Sep 2. PMID 31478089
- [Derived] Duan H, Moradi F, Davidzon GA, Liang T, Song H, Loening AM, Vasanawala S, Srinivas S, Brooks JD, Hancock S, Iagaru A. 68Ga-RM2 PET-MRI versus MRI alone for evaluation of patients with biochemical recurrence of prostate cancer: a single-centre, single-arm, phase 2/3 imaging trial. Lancet Oncol. 2024 Apr;25(4):501-508. doi: 10.1016/S1470-2045(24)00069-X. Epub 2024 Feb 26. PMID 38423030
- [Derived] Duan H, Davidzon GA, Moradi F, Liang T, Song H, Iagaru A. Modified PROMISE criteria for standardized interpretation of gastrin-releasing peptide receptor (GRPR)-targeted PET. Eur J Nucl Med Mol Imaging. 2023 Nov;50(13):4087-4095. doi: 10.1007/s00259-023-06385-z. Epub 2023 Aug 9. PMID 37555901
- [Derived] Duan H, Baratto L, Hatami N, Liang T, Levin CS, Khalighi MM, Iagaru A. Reduced Acquisition Time per Bed Position for PET/MRI Using 68Ga-RM2 or 68Ga-PSMA-11 in Patients With Prostate Cancer: A Retrospective Analysis. AJR Am J Roentgenol. 2022 Feb;218(2):333-340. doi: 10.2214/AJR.21.25961. Epub 2021 Aug 18. PMID 34406051

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (68Ga-RM2 PET/MRI)
Started | 122
Completed | 121
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (68Ga-RM2 PET/MRI)
Number analyzed (Participants) | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 85
Age, Continuous [Median (Standard Deviation); unit: years] | 68.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 113
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 98
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Tumor Lesions Detected by 68Ga-RM2 MRI vs 68Ga-RM2 PET/MRI
Description: Diagnostic performance of 68Ga-RM2 as a contrast imaging label will be assessed by magnetic resonance imaging (MRI) alone, or as a combined scan with positron emission tomography (PET, collectively PET/MRI). The outcome is reported as the number of tumor lesions detected with MRI alone, or with the combination PET/MRI scan, a number without dispersion.
Time Frame: 1 day
Measure: Number; unit: number of tumor lesions
Arm/Group | Diagnostic (68Ga-RM2 PET/MRI)
Number analyzed (Participants) | 121
number of tumor lesions
  MRI scan | 92
  PET/MRI scan | 127

2. Primary Outcome: Sensitivity of MRI Alone vs PET/MRI
Description: Sensitivity is the ability of a test to correctly identify patients who have the prostate cancer, ie, how well 68Ga-RM2 MRI vs 68Ga-RM2 PET/MRI correctly detects patients who truly have prostate cancer. Sensitivity is defined as [TP/(TP+FN)], where TP=true-positive, and FN=false-negative. The outcome is a percentage number with 95% confidence interval (95% CI). A higher % value means a greater probability that an imaging target identified as cancerous is confirmed by histology to be cancerous, and a lower % means reduced confidence in that result.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Diagnostic (68Ga-RM2 PET/MRI)
Number analyzed (Participants) | 121
percentage
  MRI scan | 48.2 [37.3 to 59.3]
  PET/MRI scan | 91.8 [83.8 to 96.6]

3. Primary Outcome: Specificity of MR Alone vs PET/MRI
Description: Specificity is the ability of a test to correctly identify patients who do not have the prostate cancer, ie, how well 68Ga-RM2 MRI vs 68Ga-RM2 PET/MRI correctly detects patients who do not have prostate cancer (does not falsely return a positive result). Specificity is defined as [TN/(TN+FP)], where TN=true-negative, and FP=false-positive. The outcome is a percentage number with 95% confidence interval (95% CI). A higher % value means a greater probability that an imaging target identified as non-cancerous is confirmed by histology to be non-cancerous, and a lower % means reduced confidence in that result.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Diagnostic (68Ga-RM2 PET/MRI)
Number analyzed (Participants) | 121
percentage of participants
  MRI alone | 97.2 [66.1 to 99.8]
  PET/MRI scan | 88.9 [73.9 to 96.9]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Diagnostic (68Ga-RM2 PET/MRI)
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 0/122
Other Adverse Events (participants affected / at risk) | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT02624518/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT02624518/ICF_001.pdf